CLINICAL TRIAL: NCT03045367
Title: Mid-term Clinical Assessment and Correlation Between Metamorphopsia, Visual Acuity and Foveal Thickness in Idiopathic Epiretinal Membrane and Cataract Surgery
Brief Title: Mid-term Evaluation of Metamorphopsia in Epiretinal Membrane Surgery
Status: Completed | Type: Observational
Sponsor: Clinica Oculistica dell'Università di Torino (Other)
Responsible Party: Principal Investigator, Marco DAL VECCHIO, MD, Medical Doctor, Clinica Oculistica dell'Università di Torino
Other Study IDs: CS/526
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Epiretinal Membrane; Cataract Senile
Keywords: Metamorphopsia; Epiretinal membrane; Vitrectomy
MeSH Terms: conditions — Epiretinal Membrane; Vision Disorders | interventions — Phacoemulsification; Lens Implantation, Intraocular; Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatients: Phacoemulsification, intraocular lens implant, vitrectomy.
  Interventions: Procedure: Phacoemulsification, intraocular lens implant, vitrectomy.

INTERVENTIONS:
Procedure: Phacoemulsification, intraocular lens implant, vitrectomy. — Cataract extraction, intraocular lens implant, vitrectomy, epiretinal membrane and inner limiting retinal membrane peeling.

SUMMARY:
This study evaluates the safety and efficacy simultaneous, trans-conjunctival, 25-Gauge vitrectomy and phacoemulsification with intraocular lens implant in patients with metamorphopsia and visual impairment due to idiopathic epiretinal membrane and cataract. All 30 patients recruited underwent complete ocular examination, visual acuity measurement with ETDRS, metamorphopsia assessment with M-Charts and Metamorphometry® and foveal thickness evaluation by sd-OCT preoperatively, at 30, 90, 180 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* age > 55 years
* visual acuity ≤ 20/40
* idiopathic epiretinal membrane
* cataract
* Amsler test positive for metamorphopsia.

Exclusion Criteria:

* previous ocular interventions
* other ocular diseases.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient of all gender, with complain of visual impairment and distortion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Metamorphopsia | Change in metamorphopsia from baseline at 180 days.
  Change in spatial degree of distortion perception
Visual Acuity | Change in visual acuity from baseline at 180 days
  Change in LogMAR visual acuity
Area of central scotoma | Change in area of central scotoma from baseline at 180 days
  Change in area, in square pixel, of central scotoma
Central fovea thickness | Change in fovea thickness from baseline at 180 days
  Change in fovea thickness in µm at the Sd OCT

IPD SHARING:
Plan to Share IPD: Undecided